CLINICAL TRIAL: NCT02079376
Title: The DIAMOND® for the Treatment of Type 2 Diabetes: Can Blood Triglycerides Level be the Predictor for Therapy Efficiency A Multicentre, Prospective, Semi-randomized Study
Brief Title: The DIAMOND® for the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MetaCure Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC CP TAN2012-60
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low blood TG patients (Experimental): subjects with baseline blood triglyceride level ≤ 1.7 mmol/l will have intervention device (DIAMOND Implantable Pulse Generator (IPG)) programmed to deliver GCM signal including the setting of automatic eating detection parameters for a 48 weeks period.
  Interventions: Device: DIAMOND System
- High blood TG patients treated with blood TG lowering therapy (Experimental): subjects with baseline blood triglyceride level > 1.7 mmol/l will have their device programmed to deliver GCM signal including the setting of automatic eating detection parameters for a 48 weeks period and will receive fenofibrate at the dose of 160mg per day
  Interventions: Device: DIAMOND System
- High blood TG patients (Placebo Comparator): subjects with baseline blood triglyceride level > 1.7 mmol/l will have their device programmed to deliver GCM signal including the setting of automatic eating detection parameters for a 48 weeks period and will receive placebo of fenofibrate administered in the same schedule as the drug.
  Interventions: Device: DIAMOND System

INTERVENTIONS:
Device: DIAMOND System — DIAMOND Implantable Pulse Generator (IPG)

SUMMARY:
Study to evaluate the efficacy of gastric stimulation (GCM) using the DIAMOND System in the improvement of glycemic control measured by changes in HbA1c.

Relationship between blood TG level and the GCM efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 through 70 years of age
* Body mass index > 30 and < 45 (kg/m2)
* Type 2 diabetes duration of at least 6 months
* Type 2 diabetic subjects treated with oral anti-diabetic agents [Sulfonylurea, Metformin, thiazolinedione (TZD) or DPP-4 inhibitors]
* Stable anti-diabetic medications for at least 3 months prior to enrollment, six months for thiazolinedione (TZD)
* The subject has been under routine diabetes care of the investigator or another single physician that can supply a medical record for at least 6 months prior to enrollment
* HbA1c 7.3% and ≤ 9.5 % on Visit 1
* Stable HbA1c, defined as no significant change (variation ≤ 0.5%) between a historical value recorded in the subject's medical record within 3 months prior to enrollment and the HbA1c gathered on Visit 1.
* Fasting blood glucose >120 and < 350 mg/dl on Visit 1.
* Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
* Stable weight, defined as no significant weight change (variation <3%) within three months prior to enrollment as documented in the subject's medical record. For the subject treated with thiazolinedione, stable weight within six months.
* If taking theses medication, sable anti-hypertensive and lipid-lowering medication for at least one month prior to enrollment
* If subject is under anti-depressant medication the treatment needs to be stable for at least six months prior to enrollment.
* Ability and willingness to perform required study and data collection procedures and adhere to operating requirements of the DIAMOND System
* Willingness to perform at least four (3) capillary blood glucose tests per day twice a week for the duration of the study
* Willingness to refrain from using prescription, over the counter or herbal weight loss products for the duration of the trial
* Alert, mentally competent, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
* Able to provide voluntary informed consent

Exclusion Criteria:

* Insulin therapy in last 3 months
* Taking GLP-1 agonists or in the last 3 months before the enrollment
* Currently taking fibrates, nicotinamide and omega 3 fatty acids as antilipidemic treatment
* Subjects with an EF less than 35% or otherwise indicated for an ICD
* Taking medications known to affect gastric motility such as narcotics (chronic use) and anticholinergics/antispasmodics
* Experiencing severe and progressing diabetic complications (i.e. retinopathy not stabilized, nephropathy with macroalbuminuria)
* Prior wound healing problems due to staphylococcus or candida
* Diagnosed with past or current psychiatric condition that may impair his or her ability to comply with the study procedures
* Use of anti-psychotic medications
* Diagnosed with a eating disorder such as bulimia or binge eating
* Obesity due to an endocrine disorder (e.g. Cushing disease)
* Pregnant or lactating
* Diagnosed with impaired liver function (liver enzymes 3 times greater than normal)
* Any prior bariatric surgery
* Any history of pancreatitis
* Any history of peptic ulcer disease within 5 years of enrollment
* Diagnosed with gastroparesis
* Use of active medical devices (either implantable or external) such as ICD, pacemaker, drug infusion device, or neurostimulator (either implanted or worn). Subjects using an external active device who are able and willing to avoid use of the device during the study may be enrolled.
* Cardiac history that physician feels should exclude the subject from the study.
* Use of another investigator device or agent in the 30 days prior to enrollment
* A history of life-threatening disease within 5 years of enrollment
* Change in diabetic medication from between Visit 1 and Visit 3.
* Any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
improvement of HbA1c | 48 weeks
  improvement of glycemic control measured by changes in HbA1c

SECONDARY OUTCOMES:
Relationship between blood TG level and the GCM efficacy | 48 weeks
  Relationship between blood TG level and the GCM efficacy

CONTACTS AND LOCATIONS:
Locations (13):
- Epworth Research Institute, Richmond, Victoria, Australia
- Tilak Innsbruck, Innsbruck, Austria
- Greece (2):
  - "Attikon" Hospital, Athens
  - "Evgenidio " Hospital, Athens
- Italy (2):
  - Clinica Pineta Grande, Rome
  - The Università Cattolica del Sacro Cuore, Rome
- Poland (5):
  - Medical University, Bialystok
  - Medical University, Bydgoszcz
  - "Diabeta-Care", Lubin
  - Medical University, Szczecin
  - Centre for Postgraduate Medical Education (CMKP), Warsaw
- Serbia (2):
  - Klinika za digestivnu hirurgiju, Belgrade
  - Institut za pluće bolesti Vojvodine, Kamenica